CLINICAL TRIAL: NCT01438749
Title: Human Abuse Liability Study in Recreational Drug Users to Investigate the Abuse Liability Potential of RO4917838
Brief Title: A Study of The Abuse Liability Potential of RO4917838 in Recreational Drug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Double
Other Study IDs: BP25259
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: diazepam
- B (Placebo Comparator)
  Interventions: Drug: Placebo
- C (Experimental)
  Interventions: Drug: RO4917838

INTERVENTIONS:
Drug: Placebo — Single dose
  Arms: B
Drug: RO4917838 — Single doses (3 dose levels)
  Arms: C
Drug: diazepam — Single dose
  Arms: A

SUMMARY:
This randomized, placebo- and active-controlled, crossover study will evaluate the abuse liability potential of RO4917838 in recreational drug users. In a pre-study (Part 1), subjects will receive a single dose of either diazepam or placebo in an inpatient crossover design, with a wash-out period of at least 10 days between treatments. Subjects who are clearly able to distinguish the positive control from placebo will be enrolled in the main study (Part 2) and will be randomized to single oral doses of RO4917838 (3 dose levels), diazepam and placebo in a double-blind, double-dummy inpatient crossover design. Washout-periods between the 5 treatment periods in Part 2 will be at least 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers, 18 to 55 years of age inclusive
* Recreational drug abuse experience (>/= 10 times lifetime abuse of a CNS depressant, >/= 1 abuse of CNS depressant in the previous 3 months
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Main study (Part 2): Able to differentiate between diazepam and placebo

Exclusion Criteria:

* History of any significant disease or disorder
* History or current diagnosis of substance dependence (excluding caffeine and nicotine)
* Currently seeking or history of participating in treatment for substance-related disorders, including successful completion of such treatment
* Any confirmed significant allergic reactions against any drug, or multiple allergies in the judgement of the investigator
* Positive for hepatitis B, hepatitis C or HIV infection
* Pregnant or lactating women
* Participation in an investigational drug or device study within the last 30 days prior to Day 1 of the study
* Confirmed positive drug screening at screening / any Day -1 (allowed positive THC at screening and any Day -1 and positive benzodiazepine at screening only)
* Positive alcohol breath test at screening / any Day -1
* Heavy smoker (> 20 cigarettes, > 8 pipefuls or > 8 cigars per day)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Abuse potential measured by Visual analogue scales (VAS) | approximately 11 months

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 11 months
Pharmacokinetics: plasma concentrations of RO4917838 | approximately 11 months
Pharmacodynamics: Addiction Research Center Inventory (ARCI) subscales | approximately 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Salt Lake City, Utah, United States